CLINICAL TRIAL: NCT02364648
Title: Mitochondrial Oxidative Stress and Vascular Health in Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, David Edwards, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 680076-2
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Chronic Kidney Disease
Keywords: Endothelium, vascular; MitoQ; Mitochondria; Oxidative Stress; Chronic Renal Insufficiency; Cardiovascular Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitoQ (Experimental): 4 week 20mg oral daily dose of MitoQ
  Interventions: Dietary Supplement: MitoQ
- Placebo (Placebo Comparator): 4 week 20mg oral daily placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MitoQ — Mitochondria targeted antioxidant
  Arms: MitoQ
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of mitochondria derived oxidative stress on vascular function in patients with moderate to severe Chronic Kidney Disease.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) patients are at increased risk of cardiovascular disease. Endothelial dysfunction, characterized by a reduced bioavailability in nitric oxide, is an independent predictor of cardiovascular disease in CKD. Increased oxidative stress is a potential cause of endothelial dysfunction in this patient cohort. This study investigates the role that mitochondrial derived oxidative stress plays in CKD related vascular dysfunction. In a controlled, double blinded trial, Stage 3-5 CKD patients will be randomly assigned to receive a 4 week daily dose of a mitochondria targeted antioxidant (MitoQ) or a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 - 5 Chronic Kidney Disease

Exclusion Criteria:

* History of cardiovascular disease;
* Current pregnancy;
* Uncontrolled hypertension;
* Uncontrolled hyperlipidemia;
* Current hormone replacement therapy;
* Current use of tobacco products;
* Elevated liver enzymes;
* Current autoimmune disease;
* Daily use of of antioxidants >300mg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular Function, assessed by laser Doppler flowmetry coupled with microdialysis | Change from baseline at 4 weeks
  Nitric oxide mediated cutaneous microvascular dilatory response to local heating assessed by laser Doppler flowmetry coupled with microdialysis

SECONDARY OUTCOMES:
Conduit artery endothelial dependent dilation, assessed by duplex ultrasound | Change from baseline at 4 weeks
  Brachial artery flow mediated dilation assessed by duplex ultrasound
Mitochondria derived superoxide, assessed by electron paramagnetic resonance spectroscopy | Change from baseline at 4 weeks
  Plasma mitochondria superoxide assessed by electron paramagnetic resonance spectroscopy

OTHER OUTCOMES:
Endothelial cell NADPH oxidase expression | Change from baseline at 4 weeks
  NADPH oxidase expression in human endothelial cll expression
Arterial Stiffness, assessed by central blood pressure, augmentation index and carotid artery to femoral artery pulse wave velocity | Change from baseline at 4 weeks
  Central blood pressure, augmentation index and carotid artery to femoral artery pulse wave velocity
Ambulatory Blood Pressure | Change from baseline at 4 weeks
  2h hour continuous ambulatory blood pressure monitoring
Habitual Physical Activity, assessed by accelerometry | Change from baseline at 4 weeks
  Daily habitual physical activity assessed by accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Danielle L Kirkman, PhD, Principal Investigator — University of Delaware; David G Edwards, PhD, Principal Investigator — University of Delaware
Locations (1):
- Department of Kinesiology and Applied Physiology, University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided